CLINICAL TRIAL: NCT04349826
Title: Azithromycin and Cefixime Combination Versus Azithromycin Alone for the Out-patient Treatment of Clinically Suspected or Confirmed Uncomplicated Typhoid Fever in South Asia; a Randomised Controlled Trial
Brief Title: The Azithromycin and Cefixime Treatment of Typhoid in South Asia Trial (ACT-South Asia Trial)
Acronym: ACT-South Asia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: University of Oxford (Other); Medical Research Council (Other Government); Department for International Development, United Kingdom (Other Government); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25NP
Record Dates: First submitted 2020-04-06; First posted 2020-04-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Typhoid Fever
Keywords: Uncomplicated Typhoid Fever; Azithromycin; Cefixime; treatment failure
MeSH Terms: conditions — Typhoid Fever | interventions — Azithromycin; Cefixime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin+Cefixime (Active Comparator): Azithromycin 20mg/kg/day oral dose once daily (maximum 1gm/day) AND Cefixime 20-30mg/kg/day oral dose in two divided doses (maximum 400mg bd) for 7 days.
  Interventions: Drug: Azithromycin; Drug: Cefixime
- Azithromycin+placebo (Placebo Comparator): Azithromycin 20mg/kg/day oral dose once daily (Max 1gm/day) for 7 days AND Cefixime-matched placebo for 7 days.
  Interventions: Drug: Azithromycin; Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 20 mg/kg/day for 7 days
Drug: Cefixime — cefixime 20-30 mg/kg/day for 7 days
  Arms: Azithromycin+Cefixime
Drug: Placebo — cefixime-matched placebo for 7 days
  Arms: Azithromycin+placebo

SUMMARY:
Typhoid and paratyphoid (enteric) fever affects more than 11 million children and adults globally each year including 7 million in South Asia. Up to 1% of patients who get typhoid may die of the disease and, in those that survive, a prolonged period of ill health and catastrophic financial cost to the family may follow. In the last 20 years, treatment of typhoid fever with a 7-day course of a single oral antimicrobial, such as ciprofloxacin, cefixime or azithromycin, given in an out-patient setting has led to patient recovery in 4 to 6 days without the need for expensive hospitalization. Increasing antimicrobial resistance in Asia and sub-Saharan Africa, threatens the effectiveness of these treatments and increases the risk of prolonged illness and severe disease. The recent emergence of a particularly resistant typhoid strain in Pakistan, and subsequent international spread, adds urgency to this problem and Salmonella is now listed as a high (Priority 2) pathogen by world health organisation.

Treatment with combinations of antimicrobials may be more effective for treating typhoid fever and mitigate the problems of resistance. This suggestion is based on expert opinion but not backed up by good quality evidence. The ACT-South Asia study aims to compare a combination of azithromycin and cefixime with azithromycin alone in the outpatient treatment of clinically suspected and confirmed uncomplicated typhoid fever. The total recruitment will be 1500 patients across sites in Bangladesh, India, Nepal and Pakistan. A placebo (sugar pill) will be used instead of cefixime in the single drug arm so that neither the patient nor the study team know which patient is receiving which treatment.Investigators will assess whether treatment outcomes are better with the combination after one week of treatment and at one and three month follow-up. Both antimicrobials are widely used and have excellent safety profiles. If the combination treatment is better than the single antibiotic treatment, this will be an important result for patients across South Asia and other typhoid endemic areas. This study will additionally investigate the financial implications for families and health system.

ELIGIBILITY:
Inclusion Criteria:

* A history of fever at presentation for ≥ 72 hours and a documented fever (≥37.5oC (axillary) or ≥38oC (oral))
* Age ≥ 2 years (and ≥ 10kg) to 65 years
* No clear focus of infection on initial clinical evaluation
* Malaria rapid Diagnostic test( RDT) negative; dengue nonstructural protein(NS) 1 RDT negative; scrub typhus RDT negative; c-reactive protein(CRP) rapid test ≥10 mg/L
* Able to take oral treatment
* Able to attend for follow-up and can be contacted by telephone
* Written fully informed consent to participate in the study including assent for children in addition to parental/legal guardian consent.

Exclusion Criteria:

* History of fever for >14 days
* Pregnant or positive pregnancy test or breast-feeding
* Presence of clinical symptoms or signs indicating a focal infection such as pneumonia; urinary infection, meningitis, eschar
* Obtundation, haemodynamic shock, visible jaundice, gastrointestinal bleeding or any signs of severe disease that may require immediate hospitalisation
* Being treated for TB or HIV or severe acute malnutrition
* Patients with cardiac disease
* Patient requiring intravenous antibiotics for any reason
* Previous history of hypersensitivity to any of the treatment options
* Either of the trial drugs are contraindicated for any reason (e.g. drug interactions)
* Has received azithromycin or cefixime in the last five days
* Receiving another antimicrobial and responding clinically to the treatment as judged by the attending clinician.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2150 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Failure | Within 28 days of treatment initiation
  A composite outcome of treatment failure by the 28th day after the initiation of treatment will be defined by either of the following events: 1.Clinical failure: persistence of fever on day 7 (168 h) post treatment initiation OR The need for rescue treatment as judged by the Trial Clinician OR The development of any complication (e.g., clinically significant bleeding, fall in the Glasgow Coma Scale score, perforation of the gastrointestinal tract) OR Syndromic enteric fever relapse within 28 days of initiation of treatment. 2.Microbiological failure: a positive blood-culture for S. Typhi or S. Paratyphi on day 7 of treatment regardless of the presence of fever (microbiological failure) OR blood culture-confirmed typhoid fever relapse within 28 days of initiation of treatment.

SECONDARY OUTCOMES:
Fever clearance time (FCT) in patients in each treatment arm | at least 2 days
  The FCT will be the time from the first dose of a study drug until a temperature of < 37.5°C (axillary); < 38.0°C (oral) has been achieved
Time from onset of treatment to treatment failure | Within 28 days of treatment initiation
  The time to treatment failure will be the time from the first dose of a study drug until an event occurs defined as a treatment failure
Time from symptom onset to treatment failure | Within 28 days of treatment initiation
  The time to treatment failure will be the time from the day of the first symptom until an event occurs defined as a treatment failure
Adverse event | Within 90 days
  Adverse events will be graded (grade 3/4 adverse events, serious adverse events, adverse events of any grade leading to modification of study drug dose or interruption/early discontinuation);
faecal carriage of S.Typhi or S.Paratyphi | One and three month follow-up
  Positive culture of faeces sample for S.Typhi or S.Paratyphi
cost effectiveness of treatment | Initiation of treatment and one month follow-up visit
  The incremental cost-effectiveness ratio (ICER) will comprise of the total costs per case, real outpatient and in-patient costs, total direct and indirect costs for the family and healthcare system and health outcomes converted to Disability Adjusted Life Years (DALYs). The cost per DALY averted will be compared against multipliers of the gross domestic product/capita in each of the four countries to establish the cost-effectiveness of the combination regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Buddha Basnyat, MBBS,Msc,MD, Principal Investigator — University of Oxford
Locations (1):
- Patan Hospital, Lalitpur, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be made available to researcher and public as supporting material via open access journal and /or upon request by qualified research group.

REFERENCES:
- [Background] Butler T, Sridhar CB, Daga MK, Pathak K, Pandit RB, Khakhria R, Potkar CN, Zelasky MT, Johnson RB. Treatment of typhoid fever with azithromycin versus chloramphenicol in a randomized multicentre trial in India. J Antimicrob Chemother. 1999 Aug;44(2):243-50. doi: 10.1093/jac/44.2.243. PMID 10473232
- [Background] Chinh NT, Parry CM, Ly NT, Ha HD, Thong MX, Diep TS, Wain J, White NJ, Farrar JJ. A randomized controlled comparison of azithromycin and ofloxacin for treatment of multidrug-resistant or nalidixic acid-resistant enteric fever. Antimicrob Agents Chemother. 2000 Jul;44(7):1855-9. doi: 10.1128/AAC.44.7.1855-1859.2000. PMID 10858343
- [Result] Trivedi NA, Shah PC. A meta-analysis comparing the safety and efficacy of azithromycin over the alternate drugs used for treatment of uncomplicated enteric fever. J Postgrad Med. 2012 Apr-Jun;58(2):112-8. doi: 10.4103/0022-3859.97172. PMID 22718054
- [Result] Dolecek C, Tran TP, Nguyen NR, Le TP, Ha V, Phung QT, Doan CD, Nguyen TB, Duong TL, Luong BH, Nguyen TB, Nguyen TA, Pham ND, Mai NL, Phan VB, Vo AH, Nguyen VM, Tran TT, Tran TC, Schultsz C, Dunstan SJ, Stepniewska K, Campbell JI, To SD, Basnyat B, Nguyen VV, Nguyen VS, Nguyen TC, Tran TH, Farrar J. A multi-center randomised controlled trial of gatifloxacin versus azithromycin for the treatment of uncomplicated typhoid fever in children and adults in Vietnam. PLoS One. 2008 May 21;3(5):e2188. doi: 10.1371/journal.pone.0002188. PMID 18493312
- [Result] Parry CM, Ho VA, Phuong le T, Bay PV, Lanh MN, Tung le T, Tham NT, Wain J, Hien TT, Farrar JJ. Randomized controlled comparison of ofloxacin, azithromycin, and an ofloxacin-azithromycin combination for treatment of multidrug-resistant and nalidixic acid-resistant typhoid fever. Antimicrob Agents Chemother. 2007 Mar;51(3):819-25. doi: 10.1128/AAC.00447-06. Epub 2006 Dec 4. PMID 17145784
- [Result] Girgis NI, Butler T, Frenck RW, Sultan Y, Brown FM, Tribble D, Khakhria R. Azithromycin versus ciprofloxacin for treatment of uncomplicated typhoid fever in a randomized trial in Egypt that included patients with multidrug resistance. Antimicrob Agents Chemother. 1999 Jun;43(6):1441-4. doi: 10.1128/AAC.43.6.1441. PMID 10348767
- [Derived] Giri A, Karkey A, Dongol S, Arjyal A, Maharjan A, Veeraraghavan B, Paudyal B, Dolecek C, Gajurel D, Phuong DNT, Thanh DP, Qamar F, Kang G, Hien HV, John J, Lawson K, Wolbers M, Hossain MS, Sharifuzzaman M, Luangasanatip N, Maharjan N, Olliaro P, Rupali P, Shakya R, Shakoor S, Rijal S, Qureshi S, Baker S, Joshi S, Ahmed T, Darton T, Bao TN, Lubell Y, Kestelyn E, Thwaites G, Parry CM, Basnyat B. Azithromycin and cefixime combination versus azithromycin alone for the out-patient treatment of clinically suspected or confirmed uncomplicated typhoid fever in South Asia: a randomised controlled trial protocol. Wellcome Open Res. 2021 Nov 12;6:207. doi: 10.12688/wellcomeopenres.16801.2. eCollection 2021. PMID 35097222